CLINICAL TRIAL: NCT03601507
Title: Biomarker Modulation by Alpelisib (BYL719) in Transorally Resectable, HPV-Associated HNSCC: A Phase II Window Trial
Brief Title: Alpelisib in Treating Participants With Transorally Resectable HPV-Associated Stage I-IVA Oropharyngeal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis has chosen to withdraw support for this trial
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802258478; NCI-2018-00507 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CBYL719XUS15T (Other: Novartis); 1802258478 (Other: The University of Arizona Medical Center-University Campus); P30CA023074 (NIH)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: CDKN2A-p16 Positive; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Stage I Oropharyngeal Squamous Cell Carcinoma AJCC V7; Stage II Oropharyngeal Squamous Cell Carcinoma AJCC V7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Alpelisib) (Experimental): Participants receive Alpelisib PO QD for 14-21 days in the absence of disease progression of unacceptable toxicity and then undergo surgery. Participants may receive Alpelisib for up to 28 days if surgery is delayed.
  Interventions: Drug: Alpelisib; Other: Laboratory Biomarker Analysis; Other: Pharmacodynamic Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Alpelisib — Given PO
  Other Names: BYL719; Phosphoinositide 3-kinase Inhibitor BYL719
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies how well alpelisib works in treating participants with human papillomavirus(HPV)-associated stage I-IVA head and neck cancer that can be removed by surgery. Alpelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the preliminary efficacy of neoadjuvant Alpelisib (BYL719) in patients with transorally-resectable, HPV+ head and neck squamous cell carcinoma (HNSCC), as measured by quantitative change in tumor size (change in T) following 14-21 days of treatment.

II. To evaluate the relationship between genomic PIK3CA activation to change in T.

SECONDARY OBJECTIVES:

I. To describe the tolerability of brief neoadjuvant exposure to BYL719. II. To assess the effect of BYL719 on the tumoral Ki-67 proliferation index. III. To evaluate viral and molecular mediators of response and resistance to BYL719, including viral messenger ribonucleic acid (mRNA), E6 and E7 oncoproteins, and phosphorylated (p)HER3.

OUTLINE:

Participants receive Alpelisib orally (PO) once daily (QD) for 14-21 days in the absence of disease progression of unacceptable toxicity and then undergo surgery. Participants may receive Alpelisib for up to 28 days if surgery is delayed.

After completion of study treatment, participants are followed up for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic diagnosis of p16+ squamous cell carcinoma of oropharyngeal or unknown primary metastatic to the cervical met.
2. p16 positivity is defined as ≥70% of tumor cells demonstrating diffuse cytoplasmic and nuclear staining for p16 by immunohistochemistry in a CLIA certified pathology lab.
3. Clinical stage I-IVa p16+ oropharyngeal squamous cell carcinoma, based upon the AJCC staging manual, 7th edition.
4. No evidence of distant metastatic disease.
5. Appropriate candidate and planned for primary transoral resection and/or neck dissection.
6. ECOG performance status 0-1 at time of consent.
7. Clinically or radiologically measurable disease; the primary tumor and/or neck nodes may be measurable according to RECIST 1.1(tumor diameter ≥ 1 cm; short-axis lymph node diameter ≥ 1.5 cm) OR by caliper measurement (tumor diameter ≥ 1 cm).
8. Adequate hematologic, renal and hepatic function within 4 weeks of registration, as defined by:

   a) Absolute neutrophil count (ANC) ≥ 1,500/ul b) Creatinine ≤ 1.5 x institutional upper limit of normal (ULN). c) Bilirubin ≤ 1.5 x ULN, d) AST or ALT ≤ 2.5 x ULN. e) Fasting Serum amylase ≤ 2 × ULN f) Fasting Serum lipase ≤ ULN

   Note: A redraw is permitted within the 4 weeks for screening purposes.
9. Ability to swallow and retain oral study medication as a whole tablet
10. Have signed the written informed consent

Exclusion Criteria:

1. Prior therapy for head and neck cancer is not allowed.
2. Established diagnosis of diabetes mellitus type I or not controlled type II.
3. Known hypersensitivity to alpelisib, or to any of the excipients of alpelisib.
4. Currently documented pneumonitis (Note: The chest CT scan performed at baseline for the purpose of tumor assessment should be reviewed to confirm that there are no relevant pulmonary complications present).
5. Any of the following cardiac abnormalities:

   1. Symptomatic congestive heart failure within 12 months prior to the start of study treatment
   2. History of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy
   3. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
   4. Myocardial infarction ≤ 6 months prior to start of study treatment
   5. Unstable angina pectoris
   6. Serious uncontrolled cardiac arrhythmia
   7. History of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis prior to the start of study treatment
   8. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication. (Initiation or adjustment of antihypertensive medication(s) is allowed during screening; hypertension must be controlled prior to administering the study drug.) QTcF > 480 msec on the screening ECG (using the QTcF formula)
6. Currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed.
7. Currently receiving any of the following medications and cannot be discontinued at least 7 days prior to the start of the treatment:

   1. Medications that have a known risk to prolong the QT interval or induce Torsade de Pointes (TdP) and the treatment cannot be discontinued or switched to a different medication prior to starting treatment with BYL719 (refer to list of prohibited QT prolonging drugs provided in in Appendix 3)
   2. Herbal preparations/medications
8. Currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week prior to the start of study treatment and must have discontinued strong inhibitors before the start of treatment. Switching to a different medication prior to randomization is allowed; (Refer to Appendix 2 and 3, Tables 1 and 2) for permitted and non-permitted medications).
9. History of acute pancreatitis within1 year of screening or past medical history of chronic pancreatitis
10. Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
11. History of Stevens-Johnson-Syndrome (SJS) or Toxic Epidermal Necrolysis (TEN).
12. Known positive serology for human immunodeficiency virus (HIV)
13. Any other condition, including severe and/or uncontrolled medical conditions, that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow oral study medication as a whole tablet, social/psychological complications
14. Currently taking herbal preparations/medications and dietary supplements (except for vitamins) and unwilling to stop.
15. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
16. Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

    1. Sexually active males must use a condom during intercourse while taking BYL719 and for 1 week after the final dose of BYL719, and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
    2. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 1 week after the final dose of BYL719. Highly effective contraception is defined as either:

    i. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

ii. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study subjects, the vasectomized male partner should be the sole partner for that patient] iv. Use a combination of the following (both 1+2):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
3. Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as BYL719 may decrease the effectiveness of hormonal contraceptives.

NOTE: Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

17. Active systemic infection requiring systemic antibiotics or anti-fungals within 7 days prior to first dose of study drug.

Note: Active topical infections (for example oral thrush) do not exclude a subject even if treated with systemic antibiotics or systemic antifungals.

18. Chronic hepatitis

19. Severely impaired lung function

20. Unresolved osteonecrosis of the jaw

21. Prisoners or individuals who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricklie Julian, MD, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (1):
- The University of Arizona Medical Center-University Campus, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 out of 14 patients were accrued to the trial from March 2019 to Feb 2023. The study closed to accrual prematurely in February 2023 as the drug manufacturer, Novartis pulled support for the study. 3 patients were ineligible, 6 patients started the study.
Groups:
- Treatment (Alpelisib): Participants receive Alpelisib PO QD for 10-21 days in the absence of disease progression of unacceptable toxicity and then undergo surgery. Participants may receive Alpelisib for up to 28 days if surgery is delayed.
  Alpelisib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacodynamic Study: Correlative studies
  Therapeutic Conventional Surgery: Undergo surgery
Period: Overall Study
Arm/Group | Treatment (Alpelisib)
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.69 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Change in the Sum of Response Evaluation Criteria in Solid Tumors (RECIST) -
Description: Measurable index lesions on paired, pre-and post-treatment computed tomography scans (delta change in T) with size treated as a continuous variable. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD) is the sum of target lesions have increased by >=20% and >=5 mm from nadir; Stable disease (SD) neither sufficient shrinkage to qualify for PR not sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 6
Participants
  Stable disease | 4
  Partial response | 1
  Complete response | 0
  Progressive disease | 0
  Non-evaluable | 1

2. Primary Outcome: Percent Change in Tumor Size (Change in T) in Patients With Genomic PIK3CA Pathway Alteration (PIK3CA Mutation, Amplification, and Fluorescence in Situ Hybridization [FISH] for PTEN Loss)
Description: Will compare percent change in tumor size (change in T) in patients with genomic PIK3CA pathway alteration (PIK3CA mutation, amplification, and fluorescence in situ hybridization [FISH] for PTEN loss) versus no genomic activation.
Time Frame: Baseline up to 28 days
Population: Change in tumor size is presented here. Correlative analysis for this outcome will be completed in the upcoming months.
Measure: Median (Full Range); unit: percent change
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 5
percent change | 7.6 [0 to 33.4]

3. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Will be reported descriptively, including tabulation of toxicities according to National Cancer Institut (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: Baseline up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 6
Participants
  Diarrhea | 3
  Creatinine Increased | 1
  Acute Kidney Injury | 1
  Maculopapular rash | 2
  Hyperglycemia | 2

4. Secondary Outcome: Surgical Complications
Description: The safety of this window intervention will be reported descriptively, including tabulation of toxicities according to NCI CTCAE v.4.03, surgical complications, and length of hospital stay.
Time Frame: Baseline up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 5
Participants
  No surgical complications | 5
  Surgical complications | 0

5. Secondary Outcome: Length of Hospital Stay
Description: as for outcome 4
Time Frame: Baseline up to 28 days
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 5
days | 5.8 [3 to 9]

6. Secondary Outcome: Changes in Pre- and Post-treatment Tumor Levels of Human Papillomavirus (HPV) Messenger Ribonucleic Acid (mRNA) (Quantitative Polymerase Chain Reaction [qPCR])
Description: We hypothesize that BYL719 will reduce HPV mRNA, and this will correlate with decrease in tumor size.
Time Frame: Baseline up to 28 days
Population: Data was not collected for this outcome measure.
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in Pre- and Post-treatment Tumor Levels of E6 and E7 Oncoproteins
Description: We hypothesize that BYL719 will decrease tumoral E6 and E7 oncoprotein levels, and this will correlate with decrease in tumor size
Time Frame: Baseline up to 28 days
Population: data was not collected for this outcome measure
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 0

8. Secondary Outcome: Changes in Pre- and Post-treatment Tumor Levels of Phospho - Human Epidermal Growth Factor Receptor 3 (HER3)
Description: We hypothesize that pHER3 is a resistance mechanism for BYL719, and that pHER3 will be upregulated in non-responders.
Time Frame: Baseline up to 28 days
Population: data was not collected for this outcome measure
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 0

9. Secondary Outcome: Changes in Pre- and Post-treatment Tumor Levels of HER3/PI3K Dimers (Monogram)
Description: We hypothesize that HER3/PI3K dimerization is a resistance mechanism for BYL719, and that dimers will be upregulated in non-responders.
Time Frame: Baseline up to 28 days
Population: Data was not collected for this outcome measure
Arm/Group | Treatment (Alpelisib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from each patient from the time of their first treatment with study drug. Subjects received study drug for 10-21 days. At the 4-week follow up visit, adverse drug reactions were followed until return to baseline or stabilization. At the 4 week follow-up visit, only adverse drug reactions were documented.
Description: Only AEs meeting one of the following criteria were collected.
  * Any AE that is Grade 3 or higher, regardless of relationship to the study drug
  * Any intolerable Grade 2 AE
  * Any Grade AE resulting in holding or dose-reducing BYL719
  * Any Grade 2 laboratory or vital sign values that are deemed clinically significant by the treating investigator
  * Any Grade AE in the following categories of interest:
    * Rash
    * Diarrhea
    * Pneumonitis
    * Hyperglycemia
Arm/Group | Treatment (Alpelisib)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Alpelisib) (N=6)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
This study stopped accrual early as the investigational product (IP) manufacturer, Novartis, terminated the study stopping provision of IP. 6 out of 20 subjects were accrued, 5 of which completed study. Due to early termination with few patients, only the counts of events have been calculated and no testing was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03601507/Prot_SAP_000.pdf